CLINICAL TRIAL: NCT03559010
Title: A Multi-Center Oral Contraceptive Pill Use Trial Conducted In an OTC Naturalistic Environment (OPTION)
Brief Title: A Study of Oral Contraception Under Simulated OTC Conditions
Acronym: OPTION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated prematurely due to issues with one of the data collection systems, no impact on subject safety
Sponsor: HRA Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 151042-001
Record Dates: First submitted 2018-05-18; First posted 2018-06-15 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Contraception
Keywords: Daily birth control
MeSH Terms: interventions — Norgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Use Phase Norgestrel 0.075 mg (Experimental): Norgestrel 0.075 mg tablets to be taken orally, one tablet daily at the same time everyday for up to 16 weeks
  Interventions: Drug: Norgestrel 0.075 mg tablets

INTERVENTIONS:
Drug: Norgestrel 0.075 mg tablets — All subjects enrolled in the use phase of this open-label study will be given the opportunity to purchase and take one Norgestrel 0.075 mg tablet daily up to 16 weeks.
  Subjects will use the investigational product based on their understanding of the directions on the outer packaging called the Drug Facts Label and information inside the product packaging called the Consumer Information Leaflet.
  Other Names: Opill

SUMMARY:
This study is designed to assess whether consumers select and use norgestrel 0.075 mg, a progestin only pill for contraception, in a manner consistent with the OTC package directions in an Over-the-Counter (OTC)-like setting.

DETAILED DESCRIPTION:
Subjects will be primarily recruited via passive recruiting methods, such as in-store posters, direct mail postcards, and digital space advertising.

Respondents to advertisements will either call Clinical Research Organization (CRO) call center or visit the study website for initial screening (during which data regarding age, gender, and minimal study exclusion criteria will be collected) and scheduling of an in-person enrollment visit at a local participating research site.

During the face-to-face enrollment visit, potential subjects who meet the inclusion and exclusion criteria for the study will be given an (empty) study medication package and will be allowed as much time as they need to review the information on the outside of the entire package. Subjects will then be asked if the product is OK or not OK for them to use.

Qualified subjects then will be allowed to purchase (pharmacy sites) or be given (clinic sites) the study product.

Approximately 47 sites will be used, comprising retail pharmacy research sites and women's health clinics or adolescents' clinics.

ELIGIBILITY:
Inclusion Criteria:

-Women who are willing purchase (in the pharmacies) or be provided (in the clinics) oral contraception for their own use for the purposes of the study

Exclusion Criteria:

* Cannot read, speak and understand English
* Cannot see well enough to read information on the label

Min Age: 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2018-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Bradford, MD, MSPH, Principal Investigator — Pegus Research, Inc.
Locations (41):
- United States (41):
  - HRA Pharma Investigational site, Birmingham, Alabama
  - HRA Pharma Investigational site, Homewood, Alabama
  - HRA Pharma Investigational site, McCalla, Alabama
  - HRA Pharma Investigational site, Tucson, Arizona
  - HRA Pharma Investigational site, Downey, California
  - HRA Pharma Investigational site, La Habra, California
  - HRA Pharma Investigational site, Long Beach, California
  - HRA Pharma Investigational site, Los Angeles, California
  - HRA Pharma Investigational site, Bridgeport, Connecticut
  - HRA Pharma Investigational site, Hartford, Connecticut
  - HRA Pharma Investigational site, New Haven, Connecticut
  - HRA Pharma Investigational site, Riverview, Florida
  - HRA Pharma Investigational site, Dalton, Georgia
  - HRA Pharma Investigational site, Griffin, Georgia
  - HRA Pharma Investigational site, Catonsville, Maryland
  - HRA Pharma Investigational site, Anoka, Minnesota
  - HRA Pharma Investigational site, Elk River, Minnesota
  - HRA Pharma Investigational site, Fridley, Minnesota
  - HRA Pharma Investigational Site, Saint Francis, Minnesota
  - HRA Pharma Investigational site, Elsberry, Missouri
  - HRA Pharma Investigational site, Manchester, Missouri
  - HRA Pharma Investigational Site, Savannah, Missouri
  - HRA Pharma Investigational site, Springfield, Missouri
  - HRA Pharma Investigational site, Monroe, New Jersey
  - HRA Pharma Investigational site, Albuquerque, New Mexico
  - HRA Pharma Investigational site, Burlington, North Carolina
  - HRA Pharma Investigational Site, South Charleston, Ohio
  - HRA Pharma Investigational site, Bethlehem, Pennsylvania
  - HRA Pharma Investigational site, Clarksville, Tennessee
  - HRA Pharma Investigational site, Cleveland, Tennessee
  - HRA Pharma Investigational site, Houston, Texas
  - HRA Pharma Investigational site, Sherman, Texas
  - HRA Investigational site, Bountiful, Utah
  - HRA Pharma Investigational site, Mapleton, Utah
  - HRA Pharma Investigational site, Syracuse, Utah
  - HRA Pharma Investigational site, Montpelier, Virginia
  - HRA Pharma Investigational site, Enumclaw, Washington
  - HRA Pharma Investigational site, Kenmore, Washington
  - HRA Pharma Investigational site, Seattle, Washington
  - HRA Pharma Investigational site, Snohomish, Washington
  - HRA Pharma Investigational site, Amery, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Self-selection population: participants who accept the invitation to participate and meet study inclusion criteria, participate in a face-to-face interview at the study site, make a self-selection decision, and provide responses to all relevant medical history questions.
  Purchaser Population: responders who meet study enrollment criteria and purchase/obtain the study medication.
  Use Phase Norgestrel 0.075 mg: subjects who take at least one dose of study medication during the study.
Groups:
- Self Selection Population: Males or females at least 12 years of age who presented at a pharmacy study site in response to advertising or who presented to a clinic site seeking an oral contraceptive could be enrolled in the Self-Selection population of the study
Period: Overall Study
Arm/Group | Self Selection Population
Started | 189 (The number of participants to start a period is not equal to the number who completed previous period)
Purchaser Population | 113
Use Phase Norgestrel 0.075 mg | 109
Completed | 189
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Males or females at least 12 years of age who presented at a pharmacy study site in response to advertising or who presented to a clinic site seeking an oral contraceptive could be enrolled in the Self-Selection population of the study. Of the 189 subjects who completed the Self-Selection interview, 113 (59.8%) qualified to purchase the product and proceeded to the Use Phase. 109 of 113 purchasers reported taking at least one dose of study product (User Population). The total of subjects is 189.
Groups:
- All Participants: Males or females at least 12 years of age who presented at a pharmacy study site in response to advertising or who presented to a clinic site seeking an oral contraceptive could be enrolled in the Self-Selection population of the study.
  The total number of subjects enrolled is 189. Out of the 189 subjects, 113 were included in the Purchaser population. And in 113 subjects included in Purchaser Population, 109 were in Use Phase (Users).
Arm/Group | All Participants
Number analyzed (Participants) | 189
Age, Continuous [Median (Full Range); unit: years]
  All participants | 29.0 [15 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  All participants: Female | 188
  All participants: Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  All participants: Hispanic or Latino | 31
  All participants: Not Hispanic or Latino | 156
  All participants: Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 43
  White | 117
  More than one race | 16
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 189
Literacy using REALM test pr REALM Teen test [Count of Participants; unit: Participants] — In order to address any concerns about the ability of consumers with low literacy to follow labeled instructions, subjects had their literacy level assessed by the Rapid Estimate of Adult Literacy in Medicine, a tool to screen for below-grade reading in health care settings. Adolescent subjects (<age 18) had their literacy evaluated by use of the Rapid Estimate of Adolescent Literacy in Medicine. Min score 0, max score 66. Graded as Low Health Literacy if score is below or equal to 60. Graded as Normal Health Literacy if score at least 61.
  Participants
    Normal Literacy | 167
    Low Literacy | 21
    Litercay Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Self-selection
Description: Proportion of self-selection population who make a correct selection decision regarding use of the product Study prematuraly discontinued No Self-selection endpoint calculations were made.
Time Frame: Day One
Population: The clinical trial was terminated before data are collected. No Endpoints calculations were made
Groups:
- Purchaser Population: During the face-to-face enrollment visit, potential subjects who met the inclusion and exclusion criteria for the study were given an (empty) Opill® package and were administered the enrollment interview, which comprised (1) review of the packaging, (2) determining if the product was OK or not OK for them to use and if they would like to purchase it, (3) providing limited medical history, current medication use and demographic information, (4) assessment of literacy/reading ability, (5) informed consent, (6) enrollment pregnancy test, and (7) purchase (pharmacy sites) or dispensing (clinic sites) of the Investigational Product.
- Use Phase Norgestrel 0.075 mg: Norgestrel 0.075 mg tablets to be taken orally, one tablet daily at the same time everyday for up to 16 weeks
  Norgestrel 0.075 mg tablets: All subjects enrolled in the use phase of this open-label study will be given the opportunity to purchase and take one Norgestrel 0.075 mg tablet daily up to 16 weeks.
  Subjects will use the investigational product based on their understanding of the directions on the outer packaging called the Drug Facts Label and information inside the product packaging called the Consumer Information Leaflet.
Arm/Group | Self Selection Population | Purchaser Population | Use Phase Norgestrel 0.075 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Actual Use: Use of the Study Medication Every Day
Description: Measurement tool: electronic diary Study prematurely discontinued No Actual Use primary Endpoint calculations were made
Time Frame: Up to 16 weeks
Population: the clinical trial was terminated before data are collected. No endpoints calculations were made.
Arm/Group | Self Selection Population | Purchaser Population | Use Phase Norgestrel 0.075 mg
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Actual Use: Use of the Study Medication at the Same Time of Day
Description: Measurement tool: electronic diary Study prematurely discontinued No Actual Use endpoint calculations were made.
Time Frame: Up to 16 weeks
Population: the clinical trial was terminated before data are collected. No endpoints calculations were made.
Groups:
- Self-selection Population: Males or females at least 12 years of age who presented at a pharmacy study site in response to advertising or who presented to a clinic site seeking an oral contraceptive could be enrolled in the Self-Selection population of the study
Arm/Group | Self-selection Population | Purchaser Population | Use Phase Norgestrel 0.075 mg
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Actual Use: Use of the Study Medication Without an Extended Break or Any Break Between Packs
Description: Measurement tool: electronic diary Study prematurely discontinued No Actual Use endpoint calculations were made
Time Frame: Up to 16 weeks
Population: the clinical trial was terminated before data are collected. No endpoints calculations were made.
Arm/Group | Use Phase Norgestrel 0.075 mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Actual Use: Proportion of User Population Who do Not Use Study Medication Together With Another Form of Hormone-containing Birth Control.
Description: Proportion of user population who do not use study medication together with another form of hormone-containing birth control.
  Measurement tool: electronic diary Study prematurely discontinued No Actual Use endpoint calculations were made
Time Frame: Up to 16 weeks
Population: the clinical trial was terminated before data are collected. No endpoints calculations were made.
Arm/Group | Use Phase Norgestrel 0.075 mg
Number analyzed (Participants) | 0

6. Secondary Outcome: Actual Use: Proportion of User Population Who Report Using a Barrier Method of Contraception (or Abstaining From Intercourse) for the First 48 Hours After Starting to Use the Study Medication
Description: Proportion of user population who report using a barrier method of contraception (or abstaining from intercourse) for the first 48 hours after starting to use the study medication Measurement tool: electronic diary Study prematurely discontinued No Actual Use endpoint calculations were made
Time Frame: Up to 16 weeks
Population: the clinical trial was terminated before data are collected. No endpoints calculations were made.
Arm/Group | Use Phase Norgestrel 0.075 mg
Number analyzed (Participants) | 0

7. Secondary Outcome: Proportion of Self-selection Population Taking One of the "Ask a Doctor or Pharmacist Before Use" Products Who do Not Select, Who Select But do Not Use, or Who Report Contacting a Healthcare Provider or Pharmacist About Use of the Product
Description: Proportion of self-selection population taking one of the "ask a doctor or pharmacist before use" products who do not select, who select but do not use, or who report contacting a healthcare provider Measurement tool: phone interview Study prematurely discontinued No Self-selection endpoint calculations were made
Time Frame: Up to 16 weeks
Population: the clinical trial was terminated before data are collected. No endpoints calculations were made.
Arm/Group | Use Phase Norgestrel 0.075 mg
Number analyzed (Participants) | 0

8. Secondary Outcome: Proportion of Self-selection Population Who Report Having Liver Problems Who Either do Not Select ,Who Select But do Not Use, or Who Report Contacting a Healthcare Provider About Use of the Product.
Description: Proportion of self-selection population who report having liver problems who either do not select ,who select but do not use, or who report contacting a healthcare provider about use of the product.
  Measurement tool: phone interview Study prematurely discontinued No Self-selection endpoint calculations were made.
Time Frame: Up to 16 weeks
Population: the clinical trial was terminated before data are collected. No endpoints calculations were made.
Arm/Group | Use Phase Norgestrel 0.075 mg
Number analyzed (Participants) | 0

9. Secondary Outcome: Proportion of User Population Who Experience One of the "Talk to a Doctor" Conditions Listed Within the "When Using This Product" or "Stop Use and Ask a Doctor" Sections
Description: Proportion of user population who experience one of the "Talk to a doctor" conditions listed within the "When using this product" or "Stop use and ask a doctor" sections Measurement tool: phone interview Study prematurely discontinued No User endpoint calculations were made.
Time Frame: Up to 16 weeks
Population: the clinical trial was terminated before data are collected. No endpoints calculations were made.
Arm/Group | Use Phase Norgestrel 0.075 mg
Number analyzed (Participants) | 0

10. Secondary Outcome: Safety Population: Number of Pregnancies Reported During the Course of the Study
Description: Number of pregnancies reported during the course of the study Measurement tool: phone interview
Time Frame: Up to 16 weeks
Population: Arms are combined in the safety population. The safety population included 116 subjects who provided informed consent, 113 of whom purchased the IP and entered the use phase of the study.
Measure: Number; unit: participants
Arm/Group | Use Phase Norgestrel 0.075 mg
Number analyzed (Participants) | 116
participants | 1

ADVERSE EVENTS:
Time Frame: up to 16 weeks
Groups:
- Safety Population: Arms are combined in the safety population. The safety population included 116 subjects who provided informed consent, 113 of whom purchased the IP and entered the use phase of the study.
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/116
Serious Adverse Events (participants affected / at risk) | 4/116
Other Adverse Events (participants affected / at risk) | 28/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=116)
Exposure During Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=116)
Headache (Nervous system disorders) | 3 (3)
Migraine (Nervous system disorders) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 6 (6)
Menorrhagia (Reproductive system and breast disorders) | 8 (8)
Metrorrhagia (Reproductive system and breast disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT03559010/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT03559010/SAP_001.pdf